CLINICAL TRIAL: NCT01444586
Title: Prospective Multicentre Non-interventional Study on Compliance and Patient/Doctor Behavior of VTE Prevention in Major Orthopedic Surgery
Brief Title: Russian Non-Interventional Study on Compliance of Venous Thromboembolism (VTE)
Acronym: SOPRANO
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 16002; XA2011-01RU (Other: Company Internal)
Record Dates: First submitted 2011-09-20; First posted 2011-10-03 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee
Keywords: non-interventional; Xarelto; knee replacement; hip replecement; Russia
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — The patients will be treated according to the routine practice. All the patients meeting the criteria of inclusion and exclusion to whom administration of Xarelto is indicated are fit for participation in this non-interventional study.

SUMMARY:
This is a local, prospective, multicenter, non-interventional, observational study. Primary objective is to describe how in "real life" thromboprophylaxis is carried out after the discharge from a hospital in the patients who undergo elective knee and hip replacement and who receive Xarelto during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years old
* Elective hip or knee replacement
* Planned VTE prevention with Xarelto
* Written informed consent
* The decision for treatment type and duration is taken by the investigator and is made before inclusion into the study.

Exclusion Criteria:

* Contraindications for the use of Xarelto in accordance with the effective instruction
* Any reasons of medical and non-medical character, which in the opinion of the physician can hamper participation of the patient in NIS, including a potentially low compliance, impossibility of making the final visit due to distant place of residence of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be treated according to the routine practice. All the patients meeting the criteria of inclusion and exclusion to whom administration of Xarelto is indicated are fit for participation in this non-interventional study.
Sampling Method: Non-Probability Sample
Enrollment: 2293 (Actual)
Dates: Start 2011-10; Primary Completion 2013-08 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Real life out-patient thromboprophylaxis after arthroplasty: Share of patients who follow physician's prescriptions; true duration of out-patient thromboprophylaxis; duration of treatment interruptions; in case of switching - reasons, drug regimen. | Not more than 8 weeks

SECONDARY OUTCOMES:
Descriptive characteristics of prescription behaviour of orthopedists (VTE prevention recommended at discharge): continuation of rivaroxaban, switching to other products (name, dose, duration, efficacy control), mechanical prophylaxis, etc. | Not more than 8 weeks
Adverse event characteristics (frequency, severity, relation to VTE prevention treatment, AE treatment, AE outcome) | Not more than 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Russia